CLINICAL TRIAL: NCT07142785
Title: Clinical Evaluation of With or Without Internal Limiting Membrane Peeling for Idiopathic Epiretinal Membrane Surgery: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250974
Record Dates: First submitted 2025-07-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Epiretinal Membranes
Keywords: Idiopathic epiretinal membrane; internal limiting membrane; visual field; randomized controlled trial

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be masked to the treatment group in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal limiting membrane (ILM) peeling group (Experimental): The patients will receive standard pars plana vitrectomy with ERM peeling combined with ILM peeling within an area of 3-4 disc diameters centered on the macula.
  Interventions: Procedure: Epiretinal membrane peeling combined with internal limiting membrane peeling
- No ILM peeling group (Active Comparator): The patients will receive standard pars plana vitrectomy with only ERM peeling
  Interventions: Procedure: Epiretinal membrane peeling

INTERVENTIONS:
Procedure: Epiretinal membrane peeling — All patients will receive standard pars plana vitrectomy, followed by only epiretinal membrane peeling.
  Arms: No ILM peeling group
Procedure: Epiretinal membrane peeling combined with internal limiting membrane peeling — All patients will receive standard pars plana vitrectomy, followed by epiretinal membrane peeling and internal limiting membrane peeling.
  Arms: Internal limiting membrane (ILM) peeling group

SUMMARY:
Idiopathic epiretinal membrane (ERM) is an age-related degenerative retinal condition. One of the primary treatment approaches is vitrectomy combined with epiretinal membrane peeling. However, whether to concurrently perform internal limiting membrane (ILM) peeling remains clinically controversial. Therefore, this study aims to compare the efficacy and safety of performing versus omitting ILM peeling during idiopathic ERM surgery.

DETAILED DESCRIPTION:
Idiopathic epiretinal membrane (ERM) is an age-related degenerative retinal condition. Its pathological hallmark is the formation of a fibrocellular membrane in the macular region, which can lead to retinal structural distortion and visual impairment. Epidemiological studies indicate that ERM is age-related, occurs more frequently unilaterally, and shows a positive correlation with advancing age, with incidence rates of 2% to 20% in individuals aged 50 to 70 years. The severity primarily depends on the location and thickness of the membrane and the presence of macular pseudoholes, manifesting as symptoms including visual field distortion (metamorphopsia), micropsia, and central vision loss. Studies suggest that ERM patients experiencing progressive visual decline, best-corrected visual acuity (BCVA) ≤ 0.6, or severe metamorphopsia require surgical intervention. There remains a lack of high-quality prospective RCTs evaluating the therapeutic outcomes of vitrectomy combined with ERM peeling with or without ILM peeling in idiopathic ERM patients. Therefore, this study aims to compare the efficacy and safety of performing versus omitting ILM peeling during idiopathic ERM surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years presenting to our hospital within the study period.
* Patients diagnosed with idiopathic epiretinal membrane (ERM) based on examination.
* Patients with best-corrected visual acuity (BCVA) ≤ 0.6 or the presence of metamorphopsia.

Exclusion Criteria:

* Patients with secondary ERM identified during preoperative evaluation (e.g., secondary to retinal vein occlusion).
* Patients with concomitant ocular diseases affecting the macula, such as macular degeneration, macular schisis, or macular atrophy.
* Patients with a history of ocular trauma or previous ocular surgery (except for cataract surgery).
* Patients with severe systemic diseases contraindicated for surgery.
* Patients with poor compliance or concomitant psychiatric disorders.
* Patients who participated in other clinical trials during the follow-up period or who were lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean deviation (MD) value | 6 months postoperatively
  mean deviation (MD) value from postoperative Humphrey visual field testing.

SECONDARY OUTCOMES:
Visual acuity | 6 months postoperatively
  uncorrected and corrected distance visual acuity
Ganglion cell complex | 6 months postoperatively
  Ganglion cell complex parameters on macular OCT
Recurrence rate | 12 months postoperatively
  Recurrence rate of ERM

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Center of the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No